CLINICAL TRIAL: NCT02480608
Title: Treatment of CML Patients With Imatinib and Hydroxyurea
Brief Title: Treatment of CML Patients With Imatinib and Hydroxyurea (CML2004)
Acronym: CML2004
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Thoralf Lange, Prof. Dr. med. Thoralf Lange, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 68
Record Dates: First submitted 2015-06-10; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination Imatinib + Hydroxyurea (Experimental): Patients who meet the inclusion criteria will be started on 400 mg Imatinib daily. In part 1 of the protocol, the dose of HU will be increased by 500 mg at 3-weekly intervals until the maximal tolerated dose has been reached. In part 2 of the study, patients will be randomized to receive either the combination or Imatinib monotherapy.
  Interventions: Drug: Imatinib; Drug: Hydroxyurea
- monotherapy Imatinib (Active Comparator): Imatinib monotherapy
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib
Drug: Hydroxyurea
  Arms: combination Imatinib + Hydroxyurea

SUMMARY:
The study will test the tolerability and efficacy of the combination therapy Imatinib/Hydroxyurea (HU) in patients with chronic myeloid leukemia (CML) in first chronic phase (CP1) newly diagnosted or failing interferon-based therapy.

DETAILED DESCRIPTION:
The protocol consists of a part 1, a phase I study that will enrol 20 patients, with the goal to determine the safety of the combination as well as the maximal tolerated dose. If the toxicity of the combination is acceptable, up to 200 more patients may be recruited and randomized to receive either Imatinib/HU or Imatinib alone (part 2).

Patients who meet the inclusion criteria will be started on 400 mg Imatinib daily. In part 1 of the protocol, the dose of HU will be increased by 500 mg at 3-weekly intervals until the maximal tolerated dose has been reached. In part 2 of the study, patients will be randomized to receive either the combination or Imatinib monotherapy.

Hematological and cytogenetic response will be evaluated at 3-months intervals during the first year, and at 6 months' intervals thereafter. Primary endpoints for part 1 are dose-limiting toxicity and maximal tolerated dose. Primary endpoints for part 2 are the rates of major and complete molecular response at 6, 12 and 18 months, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Ph-positive CML in CP1, newly diagnosed or resistant (hematologic or cytogenetic) or intolerant to interferon-based therapy
2. Age ≥ 18 years
3. Negative pregnancy test
4. Low- and intermediate risk patients younger than 45 with an HLA (Human Leukocyte Antigen) -matched sibling donor and medically fit to undergo allografting should be included only after they have been adequately counselled about the potential risk (of disease progression) associated with delaying the allograft
5. Informed consent

Exclusion Criteria:

1. Objective signs of disease progression beyond CP1 defined as

   * bone marrow or peripheral blood blasts > 15% and/or
   * blasts + promyelocytes ≥ 30% and/or
   * peripheral blood basophils ≥ 20% and/or
   * platelets < 100/nl and/or
   * chromosomal abnormalities in addition to the Ph chromosome
2. Findings suggestive of extramedullary involvement
3. Any severe and uncontrolled medical condition
4. Previous treatment with Imatinib (only part 2 of the study)
5. History of non-compliance
6. Simultaneous inclusion in other studies

Important note: previous treatment with Imatinib only is not an exclusion criterion for part 1 of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2004-04; Primary Completion 2011-08 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
number of participants with complete molecular response as a measure of efficacy | 18 months
  complete molecular response is achieved if BCR-ABL (breakpoint cluster region-Abelson murine leukemia) transcripts became undetectable

REFERENCES:
- [Derived] Lange T, Niederwieser C, Gil A, Krahl R, von Grunhagen U, Al-Ali HK, Jentsch-Ullrich K, Spohn C, Lakner V, Assmann M, Junghanss C, Cross M, Hehlmann R, Deininger M, Pfirrmann M, Niederwieser D. No advantage of Imatinib in combination with hydroxyurea over Imatinib monotherapy: a study of the East German Study Group (OSHO) and the German CML study group. Leuk Lymphoma. 2020 Dec;61(12):2821-2830. doi: 10.1080/10428194.2020.1786556. Epub 2020 Jul 16. PMID 32672489